CLINICAL TRIAL: NCT02162472
Title: Videocapillaroscopy Assessment During Systemic Agent Therapy in Patients With Psoriasis
Brief Title: Videocapillaroscopy Assessment During Systemic Agent Therapy in Psoriasis
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Principal Investigator, Joaquin Brieva, Associate Professor, Northwestern University
Other Study IDs: STU78102
Record Dates: First submitted 2014-06-10; First posted 2014-06-12 (Estimated); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Psoriasis
Keywords: videocapillaroscopy, psoriasis, systemic agent
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Adalimumab: Subjects will receive adalimumab as standard of care for psoriasis
- Methotrexate: Subjects will receive methotrexate as standard of care for psoriasis

SUMMARY:
The aim of this study is to determine if videocapillaroscopy could be used as an objective and reliable method to assess psoriasis severity and to document improvement during treatment by measuring changes in vascular features.

DETAILED DESCRIPTION:
This is a single-center, prospective, observational study that will recruit subjects from Northwestern University to examine the degree of improvement of psoriatic plaques during systemic therapy treatment. Thirty patients with a confirmed diagnosis of "active" psoriasis treated with a single systemic agent will be recruited from the Northwestern Medical Faculty Foundation Dermatology clinic. The study population will include 15 patients receiving adalimumab and 15 patients receiving methotrexate.

Eight visits will be completed for each subject: visit 0 (baseline) and visits 1-8 (week 2, 4, 6, 8, 12, 16 and 24). At the baseline visit, after informed consent is obtained, a capillaroscopic examination will be performed to assess for evidence of characteristic vascular alterations. If such changes are present, the remainder of the baseline visit will be completed. This includes gathering personal information (age, race, gender etc.), clinical history (time of first diagnosis, presentation site, treatment used, biopsy results if previously performed, etc.) and past medical history (including current and previous medications). At each of the subsequent visits (visit 1-8), any changes to medical history and/or medications will be obtained and recorded. At each of the eight visits, a dermatologic physical examination, including PASI and PGA scores will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a clinical diagnosis of chronic active plaque psoriasis
* Subjects eligible for systemic monotherapy (oral or biologic agents).
* Subjects with evidence of characteristic vascular alterations on capillaroscopic examination.
* Subjects who are able to complete the study visits and procedures, including completion of the DLQI questionnaire.
* Subjects who are willing to have standardized digital photographs taken of 2 different target plaque lesions on the extremities.
* Subjects who are willing to have videocapillaroscopic photographs taken of 2 different target plaque lesions as well as of 2 areas of uninvolved skin on the extremities.
* Subjects who have had a "4 week" washout period if they have recently changed systemic psoriatic therapy.

Exclusion Criteria:

* Those who do not fit the inclusion criteria.
* Subjects who are unable to understand the protocol or give informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thirty patients with a confirmed diagnosis of "active" psoriasis treated with a single systemic agent will be recruited from the Northwestern Medical Faculty Foundation Dermatology clinic. The study population will include 15 patients receiving adalimumab and 15 patients receiving methotrexate.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2015-07; Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Videocapillaroscopy assessment in psoriasis | Week 0, 2, 4, 6, 8, 12, 16 and 24
  The primary objective is to determine if videocapillaroscopy could be used as an objective and reliable method to assess psoriasis severity and to document improvement during treatment by measuring changes in vascular features.

CONTACTS AND LOCATIONS:
Overall Officials: Joaquin Brieva, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Department of Dermatology, Chicago, Illinois, United States